CLINICAL TRIAL: NCT02680301
Title: Comparing Efficacy of Topical Steroid Cream vs. Ointment Formulations Using Wet Dressings for Treatment of Atopic Dermatitis
Brief Title: Topical Steroid Formulation and Wet Wraps
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seton Healthcare Family (Other)
Responsible Party: Principal Investigator, Lucia Zoraida Diaz, Principal Investigator, Seton Healthcare Family
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-16-019
Record Dates: First submitted 2016-02-02; First posted 2016-02-11 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Dermatitis, Atopic
Keywords: Wet Wraps; Topical Steroid
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ointment Right/Cream Left (Other): Pt. will use 0.1% triamcinolone OINTMENT with wet-wrap dressing on right side and 0.1% triamcinolone CREAM with wet-wrap dressing on left side of bilateral flare of atopic dermatitis twice daily as instructed.
  Interventions: Drug: 0.1% triamcinolone CREAM; Drug: 0.1% triamcinolone OINTMENT
- Ointment Left/Cream Right (Other): Pt. will use 0.1% triamcinolone OINTMENT with wet-wrap dressing on left side and 0.1% triamcinolone CREAM with wet-wrap dressing on right side of bilateral flare of atopic dermatitis twice daily as instructed.
  Interventions: Drug: 0.1% triamcinolone CREAM; Drug: 0.1% triamcinolone OINTMENT

INTERVENTIONS:
Drug: 0.1% triamcinolone CREAM — Patients will be asked to apply a topical steroid in a cream formulation to one extremity using the wet wrap technique.
  Other Names: topical steroid cream
Drug: 0.1% triamcinolone OINTMENT — Patients will be asked to apply a topical steroid in a ointment formulation to one extremity using the wet wrap technique.
  Other Names: topical steroid ointment

SUMMARY:
The purpose of this study is to

1. Compare efficacy of 0.1% triamcinolone containing wet wrap as an ointment or as a cream formulation in patients with moderate to severe atopic dermatitis
2. The relative patient/subject acceptance and adherence will also be compared between the two wet wrap types

DETAILED DESCRIPTION:
In this study, the investigators will examine the effectiveness of wet wraps with topical steroids in different formulations for patients with a history of atopic dermatitis who are experiencing an acute flare. A validated clinical tool such Investigator's Global Assessment (IGA) will be used in order to assess severity of the condition as well as demonstrate the appropriateness of using wet wrap therapy as a treatment modality. IGA will measure intensity of the atopic dermatitis regarding erythema, lichenification, swelling and excoriation as well as subjective symptoms of the patient on a numeric scale. The treating clinician will be asked to rate their assessment before and after therapy.

Patients will be asked to apply a topical steroid in a cream formulation to one extremity and then apply the same topical steroid in an ointment formulation to the other using the wet wrap technique. One of the investigators or nursing staff will provide detailed instructions to the patient and parents on how to perform the wet dressing (this is already routinely done for patients initiating wet wrap therapy in the pediatric dermatology clinic). Patients will also be given a sealed and coded envelope containing instructions to apply one steroid formulation to the right extremity and the other to the left. In this manner the providers will be blinded to treatment modality during the follow-up visit. Only the research coordinator will have access to the envelope code key. An additional handout will also be provided to reinforce appropriate treatment technique. After several days (3-5) the patient will return to the dermatology clinic for a nurse visit and evaluation of any improvement of the affected areas as well as comparison of improvement of the right and left extremities. The physician investigator will examine the patient and measure improvement using the IGA. Detailed photos of the affected areas will also be taken. After a certain number of patients have enrolled in the study and completed it, the de-identified data will be examined by a statistician for comparison. Other studies evaluating the effectiveness of wet wraps have commonly had 40-50 patients enrolled which will likely be the target of this study. The statistician will compare the IGA before and after treatment on each side to allow for interpretation of the data. Stratification of data may include ages and/or severity (moderate vs severe).

Patient Oriented Eczema Measure (POEM) and/or a Quality of Life (QoL) index will also be provided to determine the patient's point of view regarding their management using validated tools. They will also be asked their opinion regarding if one side was better controlled than the other, if at all, as well as their personal preference for treatment of choice.

Compliance will be determined by weighing the medication before and after each visit and a medication calendar.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 3-17 experiencing a symmetric, bilateral flare of atopic dermatitis
2. The flares must reach a certain threshold for inclusion based on the investigator's global assessment scale

Exclusion Criteria:

1. Systemic infection or bacterial skin infections
2. Eczema herpeticum
3. Evidence of suppression of the Hypothalamic-Pituitary-Adrenal axis
4. Non-English or Non-Spanish speaking

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Diaz, MD, Principal Investigator — Seton: Dell Children's Medical Center: Specially for Childrens Dermatology
Locations (1):
- Specially for Children Dermatology, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krakowski AC, Eichenfield LF, Dohil MA. Management of atopic dermatitis in the pediatric population. Pediatrics. 2008 Oct;122(4):812-24. doi: 10.1542/peds.2007-2232. PMID 18829806
- [Background] Janmohamed SR, Oranje AP, Devillers AC, Rizopoulos D, van Praag MC, Van Gysel D, Goeteyn M, de Waard-van der Spek FB. The proactive wet-wrap method with diluted corticosteroids versus emollients in children with atopic dermatitis: a prospective, randomized, double-blind, placebo-controlled trial. J Am Acad Dermatol. 2014 Jun;70(6):1076-82. doi: 10.1016/j.jaad.2014.01.898. Epub 2014 Mar 31. PMID 24698702
- [Background] Devillers AC, Oranje AP. Efficacy and safety of 'wet-wrap' dressings as an intervention treatment in children with severe and/or refractory atopic dermatitis: a critical review of the literature. Br J Dermatol. 2006 Apr;154(4):579-85. doi: 10.1111/j.1365-2133.2006.07157.x. PMID 16536797
- [Background] Bingham LG, Noble JW, Davis MD. Wet dressings used with topical corticosteroids for pruritic dermatoses: A retrospective study. J Am Acad Dermatol. 2009 May;60(5):792-800. doi: 10.1016/j.jaad.2008.12.043. PMID 19389521
- [Background] Oranje AP, Devillers AC, Kunz B, Jones SL, DeRaeve L, Van Gysel D, de Waard-van der Spek FB, Grimalt R, Torrelo A, Stevens J, Harper J. Treatment of patients with atopic dermatitis using wet-wrap dressings with diluted steroids and/or emollients. An expert panel's opinion and review of the literature. J Eur Acad Dermatol Venereol. 2006 Nov;20(10):1277-86. doi: 10.1111/j.1468-3083.2006.01790.x. PMID 17062046
- [Background] Charman CR, Venn AJ, Williams HC. The patient-oriented eczema measure: development and initial validation of a new tool for measuring atopic eczema severity from the patients' perspective. Arch Dermatol. 2004 Dec;140(12):1513-9. doi: 10.1001/archderm.140.12.1513. PMID 15611432

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ointment Right/Cream Left | Ointment Left/Cream Right
Started | 22 | 18
Completed | 22 | 17
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ointment Right/Cream Left | Ointment Left/Cream Right | Total
Number analyzed (Participants) | 22 | 17 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 17 | 39
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.14 (3.88) | 7.29 (3.27) | 7.77 (3.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 10 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 6 | 8
  White | 13 | 11 | 24
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 17 | 39

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of 0.1% Triamcinolone Containing Wet Wrap as an Ointment or as a Cream Formulation in Patients With Moderate to Severe Atopic Dermatitis
Description: Change in atopic dermatitis based on physician global assessment scale: 0=clear; 1=almost clear; 2=mild disease; 3=moderate disease; 4=severe disease; 5- very severe disease
  Lower scores represent a better outcome.
Time Frame: 3-5 days
Population: Patients ages 3 to 17 experiencing a symmetric, bilateral flare of atopic dermatitis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cream; Ointment: Extremity that was treated with wet wraps and 0.1% triamcinolone in cream formulation
Arm/Group | Cream | Ointment
Number analyzed (Participants) | 39 | 39
units on a scale | 0.717 (0.65) | 0.589 (0.64)
Statistical Analysis 1: Comparison: Cream vs Ointment; Test type: Equivalence — Wilcoxon sign- rank test values with ranks from change in cream efficacy ratings minus change in ointment efficacy ratings; p = 0.22, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Patient Reported Efficacy
Description: Patient report of which topical steroid formulation was more effective
Time Frame: 3-5 days
Population: Patients ages 3 to 17 experiencing a symmetric, bilateral flare of atopic dermatitis.
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: All study participants
Arm/Group | All Subjects
Number analyzed (Participants) | 39
Participants
  Cream | 9
  Ointment | 16
  No Difference | 14

3. Other Pre Specified Outcome: Number of Patients Adhering to Treatment Protocol
Description: Patient-reported adherence to wet-wrap protocol. Medication logs were used to evaluate adherence to the treatment protocol for both steroid formulations. Patents were determined to be adhering to the protocol if the number of wet-wraps for each study arm (cream or ointment) were the same. Because the total number of wraps varied between patients (the protocol required 1-2 wraps per day for 3-5 days), we reviewed medication logs to determine that each patient completed an equivalent number of ointment and cream wraps.
Time Frame: 3-5 days
Population: Patients ages 3 to 17 experiencing a symmetric, bilateral flare of atopic dermatitis.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 39
Participants | 39

ADVERSE EVENTS:
Time Frame: 1 week
Groups:
- Ointement: 0.1% triamcinolone OINTMENT with wet-wrap dressing
- Cream: 0.1% triamcinolone CREAM with wet-wrap dressing
Arm/Group | Ointement | Cream
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT02680301/Prot_SAP_000.pdf